CLINICAL TRIAL: NCT00955773
Title: An Open-Label, Dose-Escalation, Phase IB II Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of the MEK Inhibitor GSK1120212 in Combination With Oral Everolimus in Subjects With Solid Tumors
Brief Title: A Study of the GSK MEK Inhibitor GSK1120212 and Everolimus in Cancer Subjects
Acronym: Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112110
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: GSK1120212, everolimus, solid tumors, pancreatic cancer, non-small lung cancer, KRAS-mutant; cancer
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms | interventions — trametinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I (Experimental): 20 to 30 solid tumor subjects will be dosed with GSK1120212 in combination with everolimus to identify Maximum Tolerated Dose. Subjects will continue on study drug until disease progression or withdraw consent.
  Interventions: Drug: GSK1120212 plus everolimus
- Group II (Experimental): 20 subjects with pancreatic cancer will receive the recommended dose identified in group I. Subjects will remain on study drug until disease progression or withdrawal from consent.
  Interventions: Drug: GSK1120212 plus everolimus
- Group III (Experimental): Approximately 40 lung cancer subjects will receive the recommended dose identified in group I. Subjects will remain on study until disease progression or withdrawal of consent.
  Interventions: Drug: GSK1120212 plus everolimus

INTERVENTIONS:
Drug: GSK1120212 plus everolimus — Dose escalation will begin at low doses of GSK1120212 and everolimus, then gradually increase in future cohorts. Dose escalation will continue until a recommended combination dose is identified. The recommended combination dose will be used to treat pancreatic and lung cancer patients in later groups in this study.

SUMMARY:
The purpose of this study is to determine the recommended dose and regimen for the orally administered MEK inhibitor GSK1120212 dosed in combination with everolimus in subjects with solid tumors. The escalation part of the study will determine the MTD. The combination will be further explored in the expansion part in subjects with metastatic pancreatic cancer. In addition, subjects with KRAS mutant non-small cell lung cancer will be enrolled.

DETAILED DESCRIPTION:
MEK112110 is a dose-escalation, open-label study to determine the recommended dose and regimen for the orally administered MEK inhibitor GSK1120212 dosed in combination with everolimus in subjects with solid tumors. This will be accomplished using a dose-escalation procedure starting at low doses of GSK1120212 and everolimus. Dose escalation will continue based on predefined parameters until the maximum tolerated dose is identified. The recommended doses and regimens will be selected based on the safety and pharmacokinetic profiles. The clinical activity of GSK1120212 dosed in combination with everolimus will be explored further in an expansion cohort consisting of 20 subjects with metastatic pancreatic cancer. In addition a substudy will be conducted in 40 subjects with KRAS-mutant non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Age 18 years old or older and able to swallow oral medication.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology (ECOG) scale for Dose Escalation Cohort. Subjects with ECOG of 2 can be enrolled for expansion cohort.
* Tumor Type criteria as listed in the protocol
* Fasting glucose < 126mg/dL
* Male subjects must agree to use one of the contraception methods listed in the protocol.
* A female subject is eligible to participate if she is of non-childbearing potential, and if she is of childbearing potential she must use protocol defined contraception methods.
* Calcium phosphate product less than or equal to 4.0 mmol2/L2 (50 mg2/dL2)
* Adequate organ system function as defined below in the protocol.

Exclusion Criteria:

* Malignancies related to HIV or solid organ transplant.
* Primary malignant brain tumors.
* Chemotherapy, radiotherapy, or immunotherapy within 28 days (or 42 days for prior nitrosoureas or mitomycin C) prior to the first dose of GSK1120212. Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity are permitted with approval of a GSK Medical Monitor if dosing of that agent is terminated at least 14 days prior to the first dose of GSK1120212.
* Use of an investigational anti-cancer drug within 28 days or 5 half-lives, whichever is shorter preceding the first dose of GSK1120212 - as long as a minimum of 14 days has passed between the last dose of the prior investigational anti-cancer drug and the first dose of GSK1120212.
* Previous treatment with an mTOR inhibitor unless approved by GSK Medical Monitor.
* Previous treatment with GSK1120212.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug, DMSO, or excipients. (To date there are no known FDA approved drugs chemically related to GSK1120212).
* Use of a prohibited medication (as defined in the protocol).
* Current use of anticoagulants (e.g. warfarin, heparin) at therapeutic levels within seven days prior to the first dose of GSK1120212. Low dose (prophylactic) low molecular weight heparin (LMWH) is permitted provided that subject's PT and PTT meet entry criteria. Subjects required therapeutic levels of LMWH must receive approval from GSK Medical Monitor and monitored appropriately as clinically indicated.
* Gastrointestinal disease predicted to interfere with absorption of an oral drug, systemic disease, major surgery, or social/psychological issues that in the opinion of investigators would jeopardize compliance with protocol.
* History of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
* Predisposing factors to RVO including uncontrolled hypertension, uncontrolled diabetes, uncontrolled hyperlipidemia, and coagulopathy.
* Visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for RVO or CSR.
* Intraocular pressure > 21mm Hg as measured by tonography.
* Glaucoma diagnosed within 1 month prior to study Day 1.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. Subjects previously treated for these conditions that are asymptomatic and off corticosteroids for at least two weeks are permitted. Subjects are not permitted to receive enzyme inducing anti-epileptic drugs (EIAEDs).
* Unresolved toxicity greater than common terminology criteria for adverse events (CTCAE) grade 1 from previous anti-cancer therapy except alopecia (if applicable) unless agreed to by a GSK Medical Monitor and the Investigator.
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks.
* QTc interval ≥ 480 msecs.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Pregnant or lactating female.
* History or active hepatitis B or C.
* History of HIV infection.
* Subjects on chronic antifungal therapy.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-08-17 (Actual); Primary Completion 2011-11-08 (Actual); Study Completion 2011-11-08 (Actual)

PRIMARY OUTCOMES:
AEs and changes in laboratory values and vital signs | 6 months
Response rate, CR + PR of GSK1120212 and everolimus in KRAS-mutant NSCLC. | 6 months

SECONDARY OUTCOMES:
GSK1120212 and everolimus PK parameters following repeat-dose (Day 15) administration of GSK1120212 and everolimus, including AUC(0-tau), Ct, Cmax, tmax, and t1/2, data permitting | 6 months
Tumor response as defined by RECIST 1.1. | 6 months
CA 19-9 levels compared to radiological response, per RECIST 1.1, over time for each pancreatic cancer subject | 6 months
Population PK parameters, oral clearance and oral volume of distribution of GSK1120212 and everolimus will be determined. Dependant upon the final compartmental model describing GSK1120212 + everolimus, add. PK may also be estimated. | 6 months
Clinical benefit response rate CR+PR+SD greater than 4mos | 6 months
Duration of response | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (2):
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
- GSK Investigational Site, Paris, France

REFERENCES:
- [Derived] Tolcher AW, Bendell JC, Papadopoulos KP, Burris HA 3rd, Patnaik A, Jones SF, Rasco D, Cox DS, Durante M, Bellew KM, Park J, Le NT, Infante JR. A phase IB trial of the oral MEK inhibitor trametinib (GSK1120212) in combination with everolimus in patients with advanced solid tumors. Ann Oncol. 2015 Jan;26(1):58-64. doi: 10.1093/annonc/mdu482. Epub 2014 Oct 24. PMID 25344362
- See also: Results for study 112110 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112110?search=study&search_terms=112110#rs